CLINICAL TRIAL: NCT00827749
Title: Contribution of Respiratory Plethysmography by Inductance and of Informatic Tool for the Study of Swallowing Disorders in Geriatrics (PRIOD)
Brief Title: Swallowing Disorders in Geriatrics Studied With Respiratory Plethysmography by Inductance
Acronym: PRIOD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Dr Alexandre Moreau-Gaudry, University Hospital of Grenoble
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DCIC 05 22
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2010-07

CONDITIONS: Swallowing Disorders
Keywords: swallowing disorders; geriatrics
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: respiratory plethysmography by inductance — contribution of respiratory plethysmography by inductance and informatic tool

SUMMARY:
The purpose of this study is to evaluate the efficiency of a novel non-invasive method for swallowing disorders detection in geriatrics.

DETAILED DESCRIPTION:
Interest: swallowing disorders exist at any age. More common among the elderly, their prevalence is estimated at between 15 and 50% of more than 60 years. Recognized today as a health problem of particular concern within this population, their pathological consequences are multiple and severe: inhalation pneumonia, often a complication of "the wrong track", was recognized in the USA in 1989, as 5th cause of death among patients aged 65, and the 3rd leading cause of death of patients over 85 years. Malnutrition facilitates infections by depression of the immune system and promotes the development of bedsores. The swallowing disorders resulting in an increase in the prevalence of dehydration, social isolation, but also an increase in mortality. Faced with such consequences, it is therefore necessary to have a reliable, non-invasive approach adapted to the fragility of the elderly to detect these disorders in order to promote preventive strategies and / or curative justified.

Originality: This work, which is part of a clinical approach uses a new method of swallowing study, described in A. Moreau-Gaudry's Medicine thesis : "Assets of the respiratory inductance plethysmography to the study of swallowing in geriatrics." The originality of this lies in the combination of Respiratory Plethysmography by inductance (RPI) to the informatic tool. The PRI allows continuous recording, thanks to a vest connected to a laptop, the patient's breathing rate. Readily available at the patient's bedside, it is non-invasive and perfectly suited to the fragility of the study population. The tool, by its automatic guarantees objectivity and reproducibility of the analysis of deglutitions from respiratory signal provided by the RPI.

ELIGIBILITY:
Inclusion Criteria:

* Patients major, consenting, cooperating.
* Person registered with the French Social Security or benefiting from an equivalent health insurance system

Exclusion Criteria:

* Patients do not qualify for inclusion pre-cited,
* Patients in a period of exclusion for other studies,
* Patients with behavioural problems that prevent them joining a clinical trial requiring prolonged collaboration (state of rest with minimal mobilization of the patient, a necessary condition to acquire a breathing rate of quality, and therefore an analysis of quality),
* Patient suffering from a nosocomial infection,
* Patient the acute stage of a condition involving the life of the latter,
* Patient insufficient breathing, oxygen, with respiratory failure poorly supported despite oxygen,
* Patient in respiratory failure decompensated
* Patient at the end of life

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Can we detect with a non-invasive, infra clinical, objective and non-traumatic tool, a patient's deglutitions from an automatic analysis of a recording of his breathing rate? | 2.5 hours

SECONDARY OUTCOMES:
Can we detect with a non-invasive, infra clinical, objective and non-traumatic tool pathological deglutitions from an automatic analysis of a recording of his breathing rate? | 2.5 hours
Can we have a test to classify patients into two groups - those without swallowing disorders and those with swallowing disorders - from an analysis of quantitative parameters relating to the analysis of the breathing rate? | 2.5 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Grenoble, Grenoble, Cedex 09, France